CLINICAL TRIAL: NCT01133041
Title: Prospective Comparison of NBI and i-Scan in Real-time Histological Prediction of Diminutive Colonic Polyps
Brief Title: Comparative Study of Postprocessing Imaging Systems for Diminutive Colonic Polyps
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Chang Kyun Lee, MD, PhD, Soon Chun Hyang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SCHCH2010L2
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2010-05

CONDITIONS: Diminutive Colon Polyp; Adenomatous Polyp; Hyperplastic Polyp; Colonoscopy
MeSH Terms: conditions — Adenomatous Polyps | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NBI observation (Experimental)
  Interventions: Other: Observation using NBI system
- i-Scan observation (Experimental)
  Interventions: Other: Observation using i-Scan system

INTERVENTIONS:
Other: Observation using NBI system — NBI system can improve the patterns of mucosal surface and vascularity of colonic polyp.
  Other Names: NBI, narrow band imaging (Olympus, Japan)
  Arms: NBI observation
Other: Observation using i-Scan system — I-Scan system can improve the patterns of mucosal surface and vascularity of colonic polyp.
  Other Names: i-Scan (Pentax, Japan)
  Arms: i-Scan observation

SUMMARY:
Several novel imaging technologies are currently used for detection and differentiation of colonic polyps during colonoscopy, such as NBI (Olympus), FICE (Fujinon), and i-Scan (Pentax).

Several previous studies have indicated that NBI without magnification can be useful for real-time differentiation of diminutive colonic neoplasias.

To date, however, there are no studies comparing NBI with other imaging systems (FICE or i-Scan) for differentiation of diminutive colonic polyps.

The study objectives are to compare the diagnostic efficacy of NBI with that of i-Scan in real-time prediction of diminutive colonic polyps.

In this prospective pilot study, diminutive colonic polyps detected during colonoscopy will be observed with conventional colonoscopy, thereafter will be observed with new imaging systems.

Sensitivity, specificity, and diagnostic accuracy of both NBI and i-Scan will be assessed by reference to histological results obtained by endoscopic biopsy or polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* screening or surveillance colonoscopy
* age over 18
* informed consent

Exclusion Criteria:

* history of inflammatory bowel diseases
* history of hereditary colorectal cancers and polyposis syndrome
* inability to give informed consent
* use of antiplatelet agent and anticoagulants
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic efficacy | about 1 year
  Sensitivity, specificity, and diagnostic accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Chang Kyun Lee, MD, PhD, Principal Investigator — Soon Chun Hyang University
Locations (1):
- Soon Chung Hyang University, Cheonan hospital, Cheonan, Choongnam, South Korea

REFERENCES:
- [Background] Rastogi A, Pondugula K, Bansal A, Wani S, Keighley J, Sugar J, Callahan P, Sharma P. Recognition of surface mucosal and vascular patterns of colon polyps by using narrow-band imaging: interobserver and intraobserver agreement and prediction of polyp histology. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):716-22. doi: 10.1016/j.gie.2008.09.058. PMID 19251016
- [Background] Rex DK. Narrow-band imaging without optical magnification for histologic analysis of colorectal polyps. Gastroenterology. 2009 Apr;136(4):1174-81. doi: 10.1053/j.gastro.2008.12.009. Epub 2008 Dec 10. PMID 19187781
- [Background] Hoffman A, Kagel C, Goetz M, Tresch A, Mudter J, Biesterfeld S, Galle PR, Neurath MF, Kiesslich R. Recognition and characterization of small colonic neoplasia with high-definition colonoscopy using i-Scan is as precise as chromoendoscopy. Dig Liver Dis. 2010 Jan;42(1):45-50. doi: 10.1016/j.dld.2009.04.005. Epub 2009 May 26. PMID 19473893
- [Derived] Lee CK, Lee SH, Hwangbo Y. Narrow-band imaging versus I-Scan for the real-time histological prediction of diminutive colonic polyps: a prospective comparative study by using the simple unified endoscopic classification. Gastrointest Endosc. 2011 Sep;74(3):603-9. doi: 10.1016/j.gie.2011.04.049. Epub 2011 Jul 18. PMID 21762907